CLINICAL TRIAL: NCT04738006
Title: Establishing Routine Preoperative Gastric Ultrasound for Patients With an Increased Aspiration Risk in a Swiss Teaching Hospital: A Prospective Observational Study.
Brief Title: Establishing Gastric Sonography in a Swiss Teaching Hospital
Status: Completed | Type: Observational
Sponsor: Kantonsspital Winterthur KSW (Other)
Responsible Party: Principal Investigator, Roman Meierhans, Principal Investigator, Kantonsspital Winterthur KSW
Other Study IDs: V2.0 - 08.01.2021
Record Dates: First submitted 2021-01-20; First posted 2021-02-04 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Gastric Ultrasound
Keywords: Teaching; Gastric Content; RSI; Aspiration; Gastric Volume; Sonography; Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preoperative gastric sonography may provide a validated, reliable, fast, and cost-efficient approach to assess aspiration risks in both elective and emergency patients. Practiced sonographers are able to perform point-of-care gastric sonography in a few minutes, thus severe delay in daily clinical practice should not be expected. Nevertheless, how this highly sensitive and specific tool should be best established in daily clinical practice is still unclear. There are no preexisting structured and validated trainings for this specific point-of-care ultrasound application. To address these issues, all patients with increased aspiration risk at the Institute of Anaesthesiology in Winterthur will be evaluated for participation during a one year recruiting period. Participants will receive a preoperative gastric ultrasound by a trained professional.

The aim of this investigation is to validate our structural training and proof the importance and effectiveness of this diagnostic tool to lay ground for improvement of anesthesiologic management and presumably patient safety in patients with an increased risk of a pulmonary aspiration.

DETAILED DESCRIPTION:
Aspiration pneumonias still exhibit a significant morbidity and mortality and are accountable for a significant part of anaesthesia-related deaths. Various diseases and especially emergency situations correlate with prolonged gastric emptying and therefore with a higher risk of pulmonary aspiration. In clinical practice the decision to perform a Rapid Sequence Induction (RSI) is mostly based on clinical and anamnestic findings. Preoperative gastric sonography may provide an objective, validated, non-invasive, reliable, fast, and cost-efficient approach to assess aspiration risks in both elective and emergency patients.

How this highly sensitive and specific tool may be best introduced and implemented in daily clinical practice or anesthesiologic guidelines remains unclear. Structured educational programmes or training recommendations for this point-of-care ultrasound application rarely exist.

Objectives:

1. Establish preoperative gastric sonography before Rapid Sequence Induction (RSI) and in patients with one or more aspiration risk factors scheduled for a advanced laryngeal mask (LMa) or regional anaesthesia at the Kantonsspital Winterthur, Department of Anaesthesiology.
2. Validation of our structured training/education by comparing sonographic estimated and directly measured gastric content.
3. Emphasize the importance and effectiveness of this diagnostic tool to improve anesthesiologic management.

At the Cantonal Hospital of Winterthur, a mid-size Swiss teaching hospital all residents and attending anaesthesiologists will receive a structured training in a period of 1 to 8 weeks before inclusion of the first patient. All participating staff will give written informed consent to participate in the study.

Tutors/experts are all expert sonographers on different modalities. They will receive a preceding training, consisting of a theoretic introduction and a course by a radiologist and abdominal sonography expert, certified by the Swiss Society for Sonography.

All included candidates will receive a structured preoperative sonography. Primary, a qualitative assessment of the gastric content should be performed in supine and right-lateral decubitus (RLD) position. In low volume states a right-lateral decubitus position (RLD) has the advantage of a gravitational shift to the antrum. That is why the investigators plan to perform the examination in both positions. If RLD position is not possible due to patient factors a half sitting or supine position can be tried. Gastric content will be classified into empty, fluid, solid or mixed. After identification, cross sectional area (CSA) will be measured and gastric content is estimated.

After placement of the routine naso- or orogastric tube (standard for RSI and LMa patients at our institute) the investigators compare the calculated and effective suctioned volume of the gastric content and analyse the difference and quality of the sonographic measurement.

No changes in or adaptions of the established clinical practice will be made for the sole purpose of this study. In exceptional cases the responsible anaesthesiologist is allowed to upgrade patients from an advanced laryngeal mask to a RSI (gold standard) after ultrasound performance to ensure patient safety. Downgrading from RSI to advanced laryngeal maks on base of the ultrasound results is not allowed.

ELIGIBILITY:
Inclusion Criteria:

* All elective in-hospital Rapid Sequence Inductions (RSI) and patients with one or more aspiration risk factors scheduled for a advanced laryngeal mask or regional anaesthesia with informed consent.
* All emergency in-hospital RSIs and patients with one or more aspiration risk factors scheduled for an advanced laryngeal mask or regional anaesthesia with informed consent graded "Notfall 1-6h, nicht vital (dringlicher Eingriff)" or, "Notfall 6-24h nicht vital (aufgeschobener dringlicher Eingriff)" according to the Swiss Society for Anaesthesiology and Resuscitation (A-QUA).

Exclusion Criteria:

* Life threatening/ time critical emergency interventions, graded followingly according to the Swiss Society for Anaesthesiology and Resuscitation (A-QUA): Notfall <1h, vital (sofortiger Eingriff notwendig)
* Known pregnancy
* Obstetric surgery
* Underage (< 18 years)
* Absence of informed consent (missing or inability to provide)
* No anaesthetist with completed structural education is available.
* Contraindications for naso- or orogastric tubes or inability to correctly place such.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Within a study period of 12 months (estimated), all elective and emergency patients scheduled for a Rapid Sequence Induction (RSI) and patients with one or more aspiration risk factors scheduled for a advanced laryngeal mask or regional anaesthesia will be screened for possible participation in this study. The indication for RSI and aspiration risk evaluation is previously determined by the responsible anaesthetist and based on patient medical history and clinical findings according to department standards.
  After evaluation of eligibility, the responsible anaesthesiologist will work through the list of inclusion and exclusion criteria. Of note, patients which are of the highest urgency where a delay is medically and ethically not acceptable, will not be included in this study. Also, patients where ability to consent is not given due to patient or circumstantial reasons, will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 2003 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Training Validation | 1 year
  Correlation of sonographic estimated gastric volume (CSA to ml) with volume aspirated (ml) through a naso- or oro-gastric tube, that was placed by routine due to the RSI or LMa procedure itself.

SECONDARY OUTCOMES:
Training Performance 1: Descriptive over all sonographies performed | 1 year
  Indirect success factors during program will be assessed as a direct PDMS (patient data management system) based feedback after each sonography in form of a questionnaire: time for examination (minutes), need of supervision (yes/no), correction of results by supervisor (yes/no), sonography difficulty (easy/medium/hard), inability to perform sonography (yes/no). Descriptive Statistics of the results including the whole study population.
Training Performance 2: over time | 1 year
  Correlation of time for examination (min), need of supervision (yes/no), correction of results corrected by supervisor (yes/no), sonography difficulty (easy/medium/hard), inability to perform sonography (yes/no) with number of examinations over time (number of sonographies), assessed over the institute (all participants) and individual learning curves. Correlation with experience in sonography, personal interest of the sonographer, job level of the examiner.
Training Performance 3: Confounders | 1 year
  Correlation of possible confounders (patient characteristics as BMI in kg/m2, American Society of Anesthesiologists (ASA) classification 1-5, patient position supine/sitting/right sided, ultrasound machine model) in Training Performance 1 and 2 analyses.
Patient population and fasting/gastric volume | 1 year
  Correlation of gastric volume (ml), fasting with time since last ingestion p.o. (h), patient characteristics as BMI (kg/m2)/ASA (1-5)/type of surgery/A-QUA and individual aspiration risk factors (as renal insufficiency, non-fasted patients, trauma, diabetes, BMI). Correlation of non-fluid CSA (cm2) with above factors and number of Aspirations in the population.
Anesthesiologic Management 1: descriptive | 1 year
  Subjective examiner rated aspiration risk (1-10) before and after sonography. Theoretical adaption of anesthesiologic management (more strict, more liberal).
Anesthesiologic Management 2: Correlation | 1 year
  Correlation of examiner rated risk and management adaption with patient and surgery factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital Winterthur, Winterthur, Canton of Zurich, Switzerland

DOCUMENTS (1):
  • Study Protocol (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT04738006/Prot_001.pdf